CLINICAL TRIAL: NCT06802705
Title: The Impact of Psychosocial Stress on Quality of Life in Saudi Arabian Patients with Alopecia Areata
Brief Title: Psychosocial Stress on QOL in Saudi Arabian Patients with Alopecia Areata
Status: Completed | Type: Observational
Sponsor: University of Jeddah (Other)
Responsible Party: Principal Investigator, Sultana Naif Kadasa, Dr, King Abdulaziz University
Other Study IDs: QOL with Alopecia Areata
Record Dates: First submitted 2025-01-07; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Hair Loss; Autoimmune Disorder; Dermatological Conditions
MeSH Terms: conditions — Alopecia Areata; Alopecia; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Psychosocial Stress on Quality of Life — Psychosocial Stress on Quality of Life in Saudi Arabian Patients with Alopecia Areata

SUMMARY:
Background: Alopecia areata (AA) is an autoimmune disorder that causes non-scaring hair loss, and common psychiatric comorbidities such as depression and anxiety are often experienced among these patients. The underlying causes of this disorder, including environmental factors, immune responses, autoimmune reactions, and genetic predisposition, are still debated. This condition affects approximately 0.2% of the global population and has no specific gender preference, with an average onset age of 33 years. This study aims to assess the psychosocial impact on quality of life in individuals with alopecia areata in Saudi Arabia Methodology: This study employed a cross-sectional questionnaire survey among Alopecia areata patients, targeting both Saudi and non-Saudi participants of both genders, from October 2023 - March 2024. The sample size is determined to be 384 participants based on a confidence level of 95%. By investigating the psychological impact of AA in Saudi Arabia.

DETAILED DESCRIPTION:
Introduction:

Hair loss is the main symptom of Alopecia areata (AA), which is caused by an autoimmune process. The pathophysiology of this disease is frequently debated; the most prevalent topics are factors related to the environment, non-specific immune responses, organ-specific autoimmune reactions, and genetic background. Furthermore, psychiatric comorbidities such as depression, anxiety, social phobia, and personality problems are very common among AA patients. Alopecia areata, which affects 0.2% of people globally, causes non-scarring hair loss. There is no obvious gender preference, and the typical age of onset is 33 years. Unpredictability exists in the disease's progression. 34-50% of patients will demonstrate spontaneous recovery 1 year after the disease's beginning, according to earlier research. According to other research, up to 80% of patients would make a full recovery after a year; however, 15-25% of patients would lose all of their body and/or head hair, and fewer than 10% of these patients would make a full recovery. Patients with dermatological conditions are far more likely to have psychiatric diseases. It has been estimated that 25% to 43% of patients visiting dermatological clinics have psychological illnesses. Studies have indicated that people with alopecia are more likely to experience psychological disorders throughout their lifespan, such as severe depression (39%) and generalized anxiety disorder (39%). Looking at the literature, research done in Makkah revealed that a considerable 79.6% of participants said that AA had a detrimental impact on one's psychological well-being. Anxiety (47.9%), depression (36.0%), and feeling criticized in front of others (63.0%) were the most prevalent psychological effects of AA. Furthermore, a study by " Abideen F" showed that in 70% of cases, the quality of life measured by the DLQI score was affected, and a history of stress was associated with 28 of the 60 patients with AA, and 17 of them suffered from psychiatric illness. Another study was done by Suchana et al (2020), aimed to investigate depression and anxiety in patients with alopecia areata, According to the study's results, anxiety and depression were both common in 75 individuals, with respective prevalence rates of 66.7% and 73.3%. Due to insignificant number of published studies that focus on the psychosocial impact of alopecia areata among patients in Saudi Arabia, Consequently, exploring this area of study is highly recommended. This study aims to assess the psychosocial impact on quality of life in individuals with alopecia areata in Saudi Arabia

Materials and Methods:

Study design: This study was a cross-sectional questionnaire survey, based on a structured questionnaire that was developed by the authors, conducted among Alopecia areata patients in Saudi Arabia.

Study setting: Participants, recruitment, and sampling procedure: This study population consisted of Alopecia areata patients in Saudi Arabia of both genders from October 2023 - March 2024.

Inclusion and Exclusion criteria:

Saudi and non-Saudi patients with Alopecia areata in Saudi Arabia who were at least 16 years old, of both sexes, and with all clinical forms of AA met the inclusion criteria. Patients who are below 16 years old and who were ineligible due to medical reasons, and those who had any concomitant chronic dermatological problems, were excluded.

Sample size:

Using the Raosoft calculator, a sample size of 384 was estimated with a confidence level of 95%. The size of the sample was calculated by using formula: n= P (1-P) * Zα 2

/ d 2with a 95 % confidence level. n: Calculated sample size Z: The z-value for the selected level of confidence (1- a) = 1.96. P: An estimated prevalence of knowledge Q: (1 - 0.50) = 50%, i.e., 0.50 D: The maximum acceptable error = 0.05. So, the calculated minimum sample size was: n = (1.96)2 X 0.50 X 0.50/ (0.05) 2 = 384.

Method for data collection and instrument (Data collection Technique and tools):

A structured questionnaire was used as a study tool. This questionnaire was developed from previous studies on the same topic, with permission obtained from the authors. The questionnaire consisted of 25 questions divided into four sections. Section 1 focused on socio-demographic characteristics and consisted of 9 questions. Section 2 assessed disease diagnosis and management approaches with 6 questions. Section 3 evaluated the psychological impact of the patients with 5 questions. Section 4 examined the quality of life of the patients with 5 questions.

In Section 1, participants were asked about their gender, age, nationality, place of residence, educational level, social status, family history of alopecia areata, sources of knowledge about alopecia areata, and type of alopecia they have. Section 2 included questions about when the disease was diagnosed, the onset of the disease, the method of diagnosis, referral to a dermatology clinic, and methods used to treat alopecia areata. Section 3 consisted of Yes/No questions and one multiple-choice question to assess the patient's feelings. Finally, Section 4 contained questions to assess the impact of alopecia areata on the patient's daily activities, such as work/school attendance, shopping habits, gardening activities, or home maintenance.

Scoring system: The authors have created a scoring system for analysis of participants response. In our survey, participants were asked about Psychosocial Stress on Quality of Life in Individuals with Alopecia areata. Each question had four valid answers. Each answer had its respective score, "Never 0, sometimes=1, usually=2, always=3". The cumulative score of the response was used to classify the participant into a risk category, "Low risk =1-6, Moderate risk =7-9, High risk =10-12".

The validated questionnaire, which was collected from a number of identical research studies and shown in the appendix, was used to evaluate Psychosocial Stress on Quality of Life in Individuals with Alopecia areata as our methodology describes.

Analyzes and entry method: Data was entered on the computer using the "Microsoft Office Excel Software" program (2016) for windows. Data was then transferred to the Statistical Package of Social Science Software (SPSS) program, version 20 (IBM SPSS Statistics for Windows, Version 20.0. Armonk, NY: IBM Corp.) to be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Saudi and non-Saudi patients with Alopecia areata in Saudi Arabia who were at least 16 years old, of both sexes, and with all clinical forms of AA met the inclusion criteria.

Exclusion Criteria:

* Patients who are below 16 years old and who were ineligible due to medical reasons, and those who had any concomitant chronic dermatological problems, were excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study population consisted of Alopecia areata patients in Saudi Arabia of both genders. Saudi and non-Saudi patients with Alopecia areata in Saudi Arabia who were at least 16 years old, of both sexes, and with all clinical forms of AA met the inclusion criteria. Patients who are below 16 years old and who were ineligible due to medical reasons, and those who had any concomitant chronic dermatological problems, were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The Impact of Psychosocial Stress on Quality of Life in Saudi Arabian Patients with Alopecia Areata | Baseline
  For this study, sociodemographic characteristics of the participants, sources of information about alopecia areata, determinants of alopecia areata, levels of psychological stress, and the potential impact of psychological stress on the quality of life of alopecia areata patients will be presented using numbers and percentages.
  The association between sociodemographic variables and the risk of psychological stress will be assessed using the chi-square test.
  The significance level for this study is chosen before data collection, and is set to be lower than 5%.

CONTACTS AND LOCATIONS:
Overall Officials: Saud Aleissa, Principal Investigator — MD FAAD, Assistant Professor, King Abdulaziz University and University Hospital, Jeddah, Saudi Arabia.
Locations (1):
- Saud Aleissa, Jeddah, Saudi Arabia

REFERENCES:
- [Background] Winnette R, Martin S, Harris N, Deal LS. Development of the Alopecia Areata Patient Priority Outcomes Instrument: A Qualitative Study. Dermatol Ther (Heidelb). 2021 Apr;11(2):599-613. doi: 10.1007/s13555-021-00508-w. Epub 2021 Mar 9. PMID 33751494
- [Background] Christensen T, Yang JS, Castelo-Soccio L. Bullying and Quality of Life in Pediatric Alopecia Areata. Skin Appendage Disord. 2017 Aug;3(3):115-118. doi: 10.1159/000466704. Epub 2017 Mar 24. PMID 28879186
- [Background] Liu LY, King BA, Craiglow BG. Alopecia areata is associated with impaired health-related quality of life: A survey of affected adults and children and their families. J Am Acad Dermatol. 2018 Sep;79(3):556-558.e1. doi: 10.1016/j.jaad.2018.01.048. Epub 2018 Feb 7. No abstract available. PMID 29425723
- [Background] Putterman E, Patel DP, Andrade G, Harfmann KL, Hogeling M, Cheng CE, Goh C, Rogers RS, Castelo-Soccio L. Severity of disease and quality of life in parents of children with alopecia areata, totalis, and universalis: A prospective, cross-sectional study. J Am Acad Dermatol. 2019 May;80(5):1389-1394. doi: 10.1016/j.jaad.2018.12.051. Epub 2019 Jan 8. PMID 30633941
- [Background] Bilgic O, Bilgic A, Bahali K, Bahali AG, Gurkan A, Yilmaz S. Psychiatric symptomatology and health-related quality of life in children and adolescents with alopecia areata. J Eur Acad Dermatol Venereol. 2014 Nov;28(11):1463-8. doi: 10.1111/jdv.12315. Epub 2013 Nov 16. PMID 24237476
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Abou-taleb DAE, Abd OH, Hameed E, Moubasher AEA. Journal of Clinical & Experimental Psychological Impact of Alopecia Areata on Egyptian Patients. 2021;12(1000568):1-4.
- [Background] Mesinkovska N, Craiglow B, Ball SG, Morrow P, Smith SG, Pierce E, Shapiro J. The Invisible Impact of a Visible Disease: Psychosocial Impact of Alopecia Areata. Dermatol Ther (Heidelb). 2023 Jul;13(7):1503-1515. doi: 10.1007/s13555-023-00941-z. Epub 2023 Jun 8. PMID 37289409
- [Background] Abideen F, Valappil AT, Mathew P, Sreenivasan A, Sridharan R. Quality of life in patients with alopecia areata attending dermatology department in a tertiary care centre - A cross-sectional study. J Pakistan Assoc Dermatologists. 2018;28(2):175-80.
- [Background] Alzubaidy BA, Banjar TA, Almaghrabi MA, Alkidaiwi SS, Basfar LM, Alzubaidy KA, Dhafar SK, Alharbi A. Evaluation of the Awareness, Beliefs, and Psychological Impact of Patients with Alopecia Areata in Makkah City, Saudi Arabia. Adv Med. 2023 May 23;2023:4286891. doi: 10.1155/2023/4286891. eCollection 2023. PMID 37260526
- [Background] Nadpara J, Tadke R, Faye A, Gawande S, Bhave S, Kirpekar V, et al. Study of anxiety in patients with moderate alopecia. Ann Indian Psychiatry. 2017;1(1):29.
- [Background] Jagtiani A, Nishal P, Jangid P, Sethi S, Dayal S, Kapoor A. Depression and suicidal ideation in patients with acne, psoriasis, and alopecia areata. J Ment Heal Hum Behav. 2017;22(1):50.
- [Background] Velez-Muniz RDC, Peralta-Pedrero ML, Jurado-Santa Cruz F, Morales-Sanchez MA. Psychological Profile and Quality of Life of Patients with Alopecia Areata. Skin Appendage Disord. 2019 Aug;5(5):293-298. doi: 10.1159/000497166. Epub 2019 Mar 20. PMID 31559253
- [Background] Toussi A, Barton VR, Le ST, Agbai ON, Kiuru M. Psychosocial and psychiatric comorbidities and health-related quality of life in alopecia areata: A systematic review. J Am Acad Dermatol. 2021 Jul;85(1):162-175. doi: 10.1016/j.jaad.2020.06.047. Epub 2020 Jun 17. PMID 32561373
- [Background] Titeca G, Goudetsidis L, Francq B, Sampogna F, Gieler U, Tomas-Aragones L, Lien L, Jemec GBE, Misery L, Szabo C, Linder D, Evers AWM, Halvorsen JA, Balieva F, Szepietowski J, Romanov D, Marron SE, Altunay IK, Finlay AY, Salek SS, Kupfer J, Dalgard FJ, Poot F. 'The psychosocial burden of alopecia areata and androgenetica': a cross-sectional multicentre study among dermatological out-patients in 13 European countries. J Eur Acad Dermatol Venereol. 2020 Feb;34(2):406-411. doi: 10.1111/jdv.15927. Epub 2019 Nov 12. PMID 31465592
- [Background] Disturbed sleep quality and increased depression scores in alopecia areata patients Aynure Oztekin, Coskun Oztekin.
- [Background] Mirza MA, Jung SJ, Sun W, Qureshi AA, Cho E. Association of depression and alopecia areata in women: A prospective study. J Dermatol. 2021 Aug;48(8):1296-1298. doi: 10.1111/1346-8138.15931. Epub 2021 Jun 14. No abstract available. PMID 34128269